CLINICAL TRIAL: NCT00569660
Title: Phase II Study of Azacitidine in Myelofibrosis
Brief Title: Ph II Study of Azacitidine in Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0033
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Results first posted 2011-03-30 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; MF; Leukemia; Azacitidine; Vidaza
MeSH Terms: conditions — Primary Myelofibrosis; Leukemia | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine (Experimental): 75 mg/m^2 Subcutaneous Daily for 7 days every 4 weeks
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m^2 subcutaneous daily for 7 days (every 4 week cycle)
  Other Names: Vidaza

SUMMARY:
The goal of this clinical research study is to learn if azacitidine can help to control MF. The safety of azacitidine in patients with Myelofibrosis (MF) will also be studied.

DETAILED DESCRIPTION:
Azacitidine is a drug that is designed to block certain genes in cancer cells whose job is to stop the function of the tumor-fighting genes. By blocking the "bad" genes, the tumor-fighting genes may be able to work better.

If you are found to be eligible to take part in this study, you will be able to begin treatment with azacitidine. You will receive azacitidine as an injection under the skin once a day for 7 days in a row. This will be repeated every 4 weeks (4 weeks equals 1 cycle). The first cycle of azacitidine will be given at M. D. Anderson, in an outpatient setting. Later cycles of treatment courses may be given at M. D. Anderson or by a cancer doctor in your community.

You may receive up to 12 cycles of treatment if you are responding well to treatment. You will be taken off study if your disease gets worse or intolerable side effects occur. Once you go off study, you will receive follow-up as is standard of care for your disease.

This is an investigational study. Azacitidine is FDA approved for the treatment of myelodysplastic syndrome. Its use in this study is experimental. A total of up to 34 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MF requiring therapy, including those previously treated and relapsed or refractory, or if newly diagnosed, with intermediate or high risk according to Lille scoring system (adverse prognostic factors are: Hemoglobin (Hb) < 10 g/dl, White Blood Cell (WBC) < 4 or > 30 x 10*9/L; risk group: 0 = low, 1 = intermediate, 2 = high).
* Performance 0-2 Eastern Cooperative Oncology Group (ECOG).
* Signed informed consent.
* Patients must have been off chemotherapy for 2 weeks prior to entering this study and have recovered from the toxic effects (grade 0-1) of that therapy. Patients are allowed to be on anagrelide and hydroxyurea to control high platelet and WBC counts for their safety.
* Serum bilirubin levels </= 1.5 times the upper limit of the normal range for the laboratory Upper Limit of of Normal(ULN). Higher levels are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis.
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels </= 2 x ULN.
* Serum creatinine levels </= 1.5 x ULN; unless related to the MF, as judged by treating physicians.
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment and should be advised to avoid becoming pregnant. Men must be advised to not father a child while receiving treatment with azacitidine. Both women of childbearing potential and men must practice effective methods of contraception (those generally accepted as standard of care measures).
* Age >/= 18.

Exclusion Criteria:

* Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known or suspected hypersensitivity to azacitidine or mannitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 6/7/05 to 4/4/08. All patients registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: The maximum accrual of 34 was met.
Period: Overall Study
Arm/Group | Azacitidine
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Azacitidine
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 22
Age Continuous [Median (Full Range); unit: years] | 67 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Clinical Response
Description: Objective Clinical Response includes Participants with Complete Response, Partial Response or Hematologic Improvement and No Response. Bone marrow aspiration and biopsy with cytogenetics every 2 to 4 courses.
Time Frame: Every 2 courses of 4 week therapy = each 8 weeks
Population: The statistical analysis for response rates determined on the intent-to-treat (ITT) populations. This is defined as all enrolled patients who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Azacitidine
Number analyzed (Participants) | 34
Participants
  Complete Response | 0
  Partial Response | 1
  Hematologic Improvement | 7
  No Response | 26

ADVERSE EVENTS:
Time Frame: 2 years 9 months
Arm/Group | Azacitidine
Serious Adverse Events (participants affected / at risk) | 17/34
Other Adverse Events (participants affected / at risk) | 10/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=34)
Hyperuricemia (Blood and lymphatic system disorders) | 2 (2)
Infection soft tissue (Infections and infestations) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2)
CNS Cerebrovascular Ischema (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-Neutropenic Fever (Infections and infestations) | 2 (2)
Neurology Intracranial Bleed (Vascular disorders) | 1 (1)
Edema (General disorders) | 1 (1)
Skin Desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Neutropenia Without Fever (Blood and lymphatic system disorders) | 2 (2)
Septic Arthritis Knee (Infections and infestations) | 1 (1)
Bladder Infection (Infections and infestations) | 1 (1)
Superficial Thrombosis (Vascular disorders) | 1 (1)
Hemorrhage Post Surgical (Vascular disorders) | 1 (1)
Aortic Aneurism (Cardiac disorders) | 1 (1)
Urosepsis Infection (Infections and infestations) | 1 (1)
Infection Laceration Knee (Infections and infestations) | 1 (1)
Gastrointestinal Hemorrhage (Vascular disorders) | 1 (1)
Gastrointestinal Infections (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine (N=34)
Neutropenia (Blood and lymphatic system disorders) | 10 (10)
Acute Renal Failure (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No